CLINICAL TRIAL: NCT01989299
Title: Ventricular Tachyarrhythmia Detection by Implantable Loop Recording in Patients With Heart Failure and Preserved Ejection Fraction (VIP-HF)
Brief Title: Ventricular Tachyarrhythmia Detection by Implantable Loop Recording in Patients With Heart Failure and Preserved Ejection Fraction
Acronym: VIP-HF
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, M. Rienstra, dr., University Medical Center Groningen
Other Study IDs: VIP-HF Registry
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Heart failure with preserved ejection fraction (HFpEF); ILR; ventricular tachyarrhythmias; Safety
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ILR implantation

SUMMARY:
Heart failure with preserved ejection fraction (HFPEF) is a large medical problem, for which no drug or device has a recommendation in current heart failure guidelines. Sudden cardiac death is suggested as the most common cause of death in HFPEF patients, although data is sparse. Use of an Implantable Loop Recorder (ILR) may be useful in patients with HFPEF to evaluate the incidence of sustained ventricular tachyarrhythmias. If ventricular tachyarrhythmias are seem frequently, treatment with an Implantable Cardioverter Defibrillator (ICD) may be an option in the future.

ELIGIBILITY:
Inclusion Criteria:

Clinical criteria:

1. Age >18 years
2. Written informed consent
3. HF with moderate to severe symptoms NYHA II or III
4. Hospitalization or emergency room visit for HF or symptom relief with diuretics within 12 months
5. Sinus rhythm or AF

Echocardiographic criteria:

1. LVEF >40%
2. Left atrial size (volume ≥34 mL/m2 or LA parasternal diameter ≥45), or left ventricular hypertrophy (septal thickness or posterior wall thickness ≥11 mm) or LV diastolic dysfunction (E/e' ≥13 or mean e' septal and lateral wall <9 cm/s).

Biomarker criteria:

1. BNP >100ng/L or NT-pro-BNP>400ng/L if sinus rhythm
2. BNP >300ng/L or NT-pro-BNP>1200ng/L if atrial fibrillation

Exclusion Criteria:

1. Patients unwilling or unable to sign informed consent
2. Patients with a pacemaker or ICD
3. Indication for ICD therapy according to the ESC guidelines
4. Life expectancy of less than one year
5. Significant coronary artery disease or myocardial infarction < 3 months
6. Complex congenital heart disease
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
The incidence of sustained ventricular tachyarrhythmias. | 2 years after ILR implantation
  To study the incidence of ventricular tachyarrhythmias in patients with HFPEF at high-risk for arrhythmic mortality.

SECONDARY OUTCOMES:
The incidence of atrial fibrillation (AF) in patients without baseline or history of AF | 2 years after ILR implantation
The rate of progression of AF in patients without baseline or history of AF | 2 years after ILR implantation
The incidence of HF hospitalizations, all cause mortality, cardiovascular mortality, and sudden cardiac death | 2 years after ILR implantation
The incidence of non-sustained ventricular tachyarrhythmias | 2 years after ILR implantation
Biomarkers (including ECG, Holter, echocardiography, CMR and blood biomarkers) for incident AF, and progression of AF in patients without baseline or history of AF | 2 years after ILR
Biomarkers (including ECG, Holter, echocardiography, CMR and blood biomarkers) of sustained ventricular tachyarrhythmias | 2 years after ILR implantation
Biomarkers (including ECG, Holter, echocardiography, CMR and blood biomarkers) of non-sustained ventricular tachyarrhythmias | 2 years after ILR implantation
Biomarkers (including echocardiography, ECG and other arrhythmogenic markers and blood biomarkers) for development of HF hospitalizations, sudden death, arrhythmic death, and all-cause mortality | 2 years after ILR implantation

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Rienstra, MD, PhD, Principal Investigator — University Medical Center Groningen; Isabelle C van Gelder, MD, PhD, Principal Investigator — University Medical Center Groningen; Alexander H Maass, MD, PhD, Principal Investigator — University Medical Center Groningen; Dirk J Veldhuisen, van, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
  - Elisabeth-TweeSteden Ziekenhuis (ETZ), Tilburg

REFERENCES:
- [Derived] van Woerden G, van Veldhuisen DJ, Manintveld OC, van Empel VPM, Willems TP, de Boer RA, Rienstra M, Westenbrink BD, Gorter TM. Epicardial Adipose Tissue and Outcome in Heart Failure With Mid-Range and Preserved Ejection Fraction. Circ Heart Fail. 2022 Mar;15(3):e009238. doi: 10.1161/CIRCHEARTFAILURE.121.009238. Epub 2021 Dec 22. PMID 34935412
- [Derived] van Veldhuisen DJ, van Woerden G, Gorter TM, van Empel VPM, Manintveld OC, Tieleman RG, Maass AH, Vernooy K, Westenbrink BD, van Gelder IC, Rienstra M. Ventricular tachyarrhythmia detection by implantable loop recording in patients with heart failure and preserved ejection fraction: the VIP-HF study. Eur J Heart Fail. 2020 Oct;22(10):1923-1929. doi: 10.1002/ejhf.1970. Epub 2020 Aug 21. PMID 32683763